CLINICAL TRIAL: NCT04679701
Title: Research Protocol for Using Confidence Socket Technology in Developing Regions: An Exploratory Study of New Techniques and Materials for Lower-limb Prosthetic Sockets
Brief Title: Using Direct Molding Socket Technology for Trans-tibial Prosthesis in Developing Regions
Status: Completed | Type: Observational
Sponsor: Amparo GmbH (Industry)
Collaborators: GDI Hub (Unknown); AT 2030 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20190425
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Transtibial Amputees

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recruited Amputees: The amputee participants will be recruited over the course of 6 months. Once a patient is recruited and has given consent, they will be fitted with a prosthesis using the Confidence Socket technology and be administered an initial survey. A follow-up meeting for one month after the fitting is scheduled. At the follow-up appointment adjustments to the prosthesis are made as needed and the patient is administered another survey.
  Interventions: Device: Amparo Confidence Socket

INTERVENTIONS:
Device: Amparo Confidence Socket — The Amparo Confidence Socket technology takes a different approach by starting with a prefabricated socket (https://www.amparo.world/confidence-socket-en). The socket is made from a moldable thermoplastic and has the attachment point pre-assembled. This prefabricated socket is essentially an "off-the-shelf" product that can be heated, then molded directly to the patient's residual limb. This removes many of the intermediate steps in traditional socket fabrication. The product's molding temperature is between 60-70 ˚C but the insulation of a silicone liner between the plastic and limb ensures safe temperatures for the patient. This process is currently used in several workshops in Europe and with approximately 50 patients currently using the product. In general, it has been shown to be safe and effective in creating below-knee prosthesis.

SUMMARY:
The study aims to understand how well CPOs and amputees can adapt to using the Amparo socket technology. CPOs at the APDK and The Cure will be trained to use the Amparo socket technology then use it with their consenting patients for a span of 7 months. Survey information will be collected along the way to assess how well the product is adapted by CPOs and patients.

DETAILED DESCRIPTION:
Objective:

The objective of the trial is to ascertain the benefits and the implications of using the Amparo socket technology within the context of two pre-existing prosthetic services in Eastern Africa.

Design:

The trial is a phase one, exploratory single group trial. 4 Certified Prosthetist Orthotists (CPOs) will be trained to use the Amparo socket technology. Over a 7-month period, 40 lower limb amputees will be recruited to participate in the study where they will be fitted with the Amparo socket technology. Follow-up after one month of using the product will help build understanding their experience with the new prosthetic leg.

There will be a beginning and end surveys and interviews with each of the 4 CPOs.

Video and written observations will be taken of both the traditional socket making method and the Confidence Socket method for comparison.

Amputee participant surveys and assessments will be collected at each fitting, and follow-up visit.

Intervention:

The intervention for the study is to introduce a new fitting method and product for lower limb prosthetic, namely the Amparo Confidence Socket consisting of the socket and liner components. All other components of the prosthesis should remain the same as what is typically used in the respective organizations.

Population:

Professionals who craft prosthesis for amputees (CPOs) and Below-knee amputees who are able to and desire to use a prosthesis who reside in Kenya.

Outcome Measures:

CPO comfort level, perceived competence, and acceptance of the Confidence Socket Technology.

Patient quality of life measure Patient mobility measures Comparative task model between traditional method and the Amparo socket technology

Duration and follow-up:

The trial will last approximately 7 months. Starting from the first introduction of the new technology until the final interview with each CPO has been completed.

ELIGIBILITY:
Inclusion Criteria:

Below-Knee amputees 18 years of or older Individuals who would normally receive prosthetic care from the respective organization Minimum of 4 weeks after amputation Able to read and communicate in English User must be able to use a passive valve suspension system with a knee sleeve (Donning the LLP with suspension system require moderate level of hand strength and dexterity)

-

Exclusion Criteria:

Users who have a known complication e.g. infection, open wounds, etc… Users who weigh more than 125kg (the max usage weight for the product) Users' residual limb cannot be longer than 25cm (MPT to stump end measurement) Users' residual limb cannot have distal circumference larger than 45cm (measured circumference with liner 4cm from end of stump)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: recruited from primary care clinic of APDK and the Cure respectively
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Trinity amputation and prosthesis scale | 1-2 months
  a psychometric assessment designed for lower limb amputees, will be used to assess quality of life, satisfaction, and adjustment level to using an LLP

SECONDARY OUTCOMES:
Amputee Mobility Predictor | 1-2 months
  an instrument that will be used to assess amputee's ability to ambulate
The L-test | 1-2 months
  a variation of the "up & go" test designed specifically for lower-limb amputees

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Barbareschi, PhD, Principal Investigator — Researcher GDI hub; Catherine Holloway, Study Director — Cofounder GDI Hub, Associate Professor UCL
Locations (2):
- Kenya (2):
  - AIC CURE International Hospital Kenya, Kijabe
  - Association for the Physically Disabled of Kenya (APDK), Mombasa

IPD SHARING:
Plan to Share IPD: No